CLINICAL TRIAL: NCT05110391
Title: Sperm Retrieval Rates by Microdissection Testicular Sperm Extraction in Non-obstructive Azoospermic Men Subjected to Gonadotropin Therapy
Brief Title: Sperm Retrieval Rates in Non-obstructive Azoospermic Men Subjected to Gonadotropin Therapy
Status: Completed | Type: Observational
Sponsor: ANDROFERT - Clinica de Andrologia e Reproducao Humana (Other)
Responsible Party: Principal Investigator, Sandro C. Esteves, Medical Director, ANDROFERT - Clinica de Andrologia e Reproducao Humana
Other Study IDs: ANDROFERT-03-20
Record Dates: First submitted 2021-09-27; First posted 2021-11-08 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Non-obstructive Azoospermia; Hormone Deficiency; Hypogonadism, Male; Male Infertility
Keywords: microdissection testicular sperm extraction; human chorionic gonadotropin; sperm retrieval rates; follicle-stimulating hormone; azoospermia; spermatogenic failure
MeSH Terms: conditions — Eunuchism; Infertility, Male; Azoospermia | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — spermatozoa
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- NOA_Treated: Hypogonadal patients with non-obstructive azoospermia who received gonadotropin therapy before sperm retrieval
  Interventions: Drug: Hormonal Therapy Agent
- NOA_Untreated: Hypogonadal patients with non-obstructive azoospermia who did not receive gonadotropin therapy before sperm retrieval

INTERVENTIONS:
Drug: Hormonal Therapy Agent — Consecutive patients with NOA and hypogonadism (defined by baseline total testosterone levels equal or below 350 ng/dL) subjected to microdissection testicular sperm extraction who received or not pre-sperm retrieval gonadotropin therapy.
  Other Names: recombinant human chorionic gonadotropin; recombinant FSH
  Groups: NOA_Treated

SUMMARY:
Azoospermia is defined as the complete absence of spermatozoa in the ejaculate. Two-thirds of azoospermic patients have non-obstructive azoospermia (NOA); the latter comprises up to 10% of infertile men overall. NOA is an untreatable testicular disorder associated with spermatogenic failure and is the most severe male infertility phenotype. Among the available surgical sperm retrieval techniques, microdissection testicular sperm extraction (micro-TESE) is the procedure of choice due to its high sperm retrieval success rates (SRR), minimal tissue extraction, and low complication rates. Even with the use of micro-TESE, the likelihood of retrieving sperm in patients with NOA remain suboptimal (40% to 60%). Hypogonadism is detected in approximately half of the patients with NOA. Given the role of intratesticular testosterone (ITT) levels for spermatogenesis, some studies have explored the clinical utility of testosterone optimization by medical therapy before sperm retrieval.

Moreover, some investigators have hypothesized that the follicle-stimulating hormone (FSH) reset might increase the expression of FSH receptors and improve Sertoli cell function. Hormonal therapy with human chorionic gonadotropin (hCG) has been shown to improve ITT production and decrease FSH levels in patients with NOA. The investigators, therefore, designed an observational cohort study aiming to evaluate whether hormone stimulation with gonadotropins (e.g., hCG alone or combined with FSH) previous to micro-TESE increases sperm retrieval rates in hypogonadal infertile men with NOA, candidates for sperm retrieval. The investigators hypothesize that optimizing ITT production and resetting FSH levels may improve spermatogenesis and successful sperm recovery.

DETAILED DESCRIPTION:
A single-center cohort study was conducted based on prospectively collected data inputted in an electronic medical record database, subsequently extracted and analyzed.

The diagnosis of NOA was based on medical history, physical examination, semen analysis, reproductive hormone measurements, genetic and imaging studies, and confirmed by histopathology.

Hypogonadism was defined based on total testosterone levels equal to or below 350 ng/dL, measured on a peripheric blood specimen taken in the morning (8:00 to 10:00 am).

Sample size calculation:

Based on existing evidence concerning SRR in patients subjected to micro-TESE with and without medical treatment to boost testosterone production, the investigators estimated a sample size of 464 participants (232 per group) to have an 80% chance of detecting, as significant at the 5% level, an increase in the primary outcome measure from 41% in the control group to 55% in the experimental group.

Statistical Analysis:

Demographic data will include patient age, BMI, infertility cause, testicular volume, reproductive hormone levels, histopathology findings, infertility duration, presence of clinical varicocele, and history of varicocele repair. Treatment variables will include type, dose, and duration of gonadotropin administration, change in reproductive hormone levels pre- vs. post-treatment, and sperm retrieval outcomes.

Continuous data will be presented as median and 25-75% interquartile range. Categorical data will be described by the number of cases and percentages. As appropriate, categorical and continuous data will be analyzed using the Pearson Chi-square and Kruskal-Wallis or Wilcoxon test. Logistic regression analyses will be conducted to examine the association between demographic and treatment covariates and the binary response 'sperm retrieval success' (yes/no). Computations will be carried out using JMP® PRO 13 and SAS 9.3 (SAS Institute, Cary, North Carolina, USA).

ELIGIBILITY:
Inclusion Criteria:

* Consecutive NOA patients with a baseline total testosterone level equal to or below 350 ng/dL who had a sperm retrieval procedure by microdissection testicular sperm extraction (micro-TESE) during the study period. Only patients with histopathology-confirmed NOA, absence of Y-chromosome microdeletion in the azoospermia factor 'a' (AZFa) and/or azoospermia factor 'b' (AZFB) region, and with a complete data record for analysis of primary and secondary outcomes were included.

Exclusion Criteria:

1. Patients subjected to sperm retrieval using percutaneous or non-microsurgical testicular biopsies and those with a history of a previous sperm retrieval attempt.
2. Patients who had used any medication with known potential gonadotoxic effects six months before enrollment and patients under gonadotropin treatment who lost follow-up.
3. Patients with NOA due to hypogonadotropic hypogonadism.
4. Patients who had any number of sperm detected in the ejaculate by routine semen analysis with centrifugation before micro-TESE, including the analysis carried out on the surgery day. The latter relates to the fact that our study is designed to include only patients with NOA confirmed by histopathology, from a specimen obtained during micro-TESE.
5. NOA patients with baseline total testosterone levels above 350 ng/dL.

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Hypogonadal patients with non-obstructive azoospermia seeking fertility.
Sampling Method: Probability Sample
Enrollment: 616 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Sperm retrieval rates | At least 3 months
  Sperm retrieval success rates by micro-TESE in men with non-obstructive azoospermia subjected or not to pre-operative hormonal stimulation

SECONDARY OUTCOMES:
Sperm retrieval rates according to hypogonadism status | At least 3 months
  Sperm retrieval success rates by micro-TESE in men with non-obstructive azoospermia subjected or not to pre-operative hormonal stimulation, according to hypogonadism categories based on baseline total testosterone levels
Sperm retrieval rates according to histopathology findings | At least 3 months
  Sperm retrieval success rates by micro-TESE in men with non-obstructive azoospermia subjected or not to pre-operative hormonal stimulation, according to testis biopsy histopathology findings
Predictive factors for sperm retrieval success | At least 3 months
  Assessment of independent co-variables affecting the binary response sperm retrieval (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Esteves, MD., PhD., Principal Investigator — ANDROFERT - Andrology and Human Reproduction Cente
Locations (1):
- Androfert, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Andrade DL, Viana MC, Esteves SC. Differential Diagnosis of Azoospermia in Men with Infertility. J Clin Med. 2021 Jul 16;10(14):3144. doi: 10.3390/jcm10143144. PMID 34300309
- [Background] Esteves SC, Prudencio C, Seol B, Verza S, Knoedler C, Agarwal A. Comparison of sperm retrieval and reproductive outcome in azoospermic men with testicular failure and obstructive azoospermia treated for infertility. Asian J Androl. 2014 Jul-Aug;16(4):602-6. doi: 10.4103/1008-682X.126015. PMID 24759580
- [Background] Hussein A, Ozgok Y, Ross L, Rao P, Niederberger C. Optimization of spermatogenesis-regulating hormones in patients with non-obstructive azoospermia and its impact on sperm retrieval: a multicentre study. BJU Int. 2013 Mar;111(3 Pt B):E110-4. doi: 10.1111/j.1464-410X.2012.11485.x. Epub 2012 Sep 7. PMID 22958644
- [Background] Reifsnyder JE, Ramasamy R, Husseini J, Schlegel PN. Role of optimizing testosterone before microdissection testicular sperm extraction in men with nonobstructive azoospermia. J Urol. 2012 Aug;188(2):532-6. doi: 10.1016/j.juro.2012.04.002. Epub 2012 Jun 15. PMID 22704105
- [Background] Achermann APP, Pereira TA, Esteves SC. Microdissection testicular sperm extraction (micro-TESE) in men with infertility due to nonobstructive azoospermia: summary of current literature. Int Urol Nephrol. 2021 Nov;53(11):2193-2210. doi: 10.1007/s11255-021-02979-4. Epub 2021 Aug 19. PMID 34410586
- [Background] Arshad MA, Majzoub A, Esteves SC. Predictors of surgical sperm retrieval in non-obstructive azoospermia: summary of current literature. Int Urol Nephrol. 2020 Nov;52(11):2015-2038. doi: 10.1007/s11255-020-02529-4. Epub 2020 Jun 9. PMID 32519242
- [Background] Laursen RJ, Elbaek HO, Povlsen BB, Lykkegaard J, Jensen KBS, Esteves SC, Humaidan P. Hormonal stimulation of spermatogenesis: a new way to treat the infertile male with non-obstructive azoospermia? Int Urol Nephrol. 2019 Mar;51(3):453-456. doi: 10.1007/s11255-019-02091-8. Epub 2019 Feb 11. No abstract available. PMID 30756283
- [Background] Esteves SC. Clinical management of infertile men with nonobstructive azoospermia. Asian J Androl. 2015 May-Jun;17(3):459-70. doi: 10.4103/1008-682X.148719. PMID 25677138
- [Background] Esteves SC. Microdissection testicular sperm extraction (micro-TESE) as a sperm acquisition method for men with nonobstructive azoospermia seeking fertility: operative and laboratory aspects. Int Braz J Urol. 2013 May-Jun;39(3):440; discussion 441. doi: 10.1590/S1677-5538.IBJU.2013.03.21. PMID 23849579
- [Background] Esteves SC, Agarwal A. Reproductive outcomes, including neonatal data, following sperm injection in men with obstructive and nonobstructive azoospermia: case series and systematic review. Clinics (Sao Paulo). 2013;68 Suppl 1(Suppl 1):141-50. doi: 10.6061/clinics/2013(sup01)16. PMID 23503964
- [Background] Tharakan T, Corona G, Foran D, Salonia A, Sofikitis N, Giwercman A, Krausz C, Yap T, Jayasena CN, Minhas S. Does hormonal therapy improve sperm retrieval rates in men with non-obstructive azoospermia: a systematic review and meta-analysis. Hum Reprod Update. 2022 Aug 25;28(5):609-628. doi: 10.1093/humupd/dmac016. PMID 35526153
- [Derived] Esteves SC, Achermann APP, Miyaoka R, Verza S Jr, Fregonesi A, Riccetto CLZ. Clinical factors impacting microdissection testicular sperm extraction success in hypogonadal men with nonobstructive azoospermia. Fertil Steril. 2024 Oct;122(4):636-647. doi: 10.1016/j.fertnstert.2024.06.013. Epub 2024 Jun 22. PMID 38909671